CLINICAL TRIAL: NCT00975065
Title: A 24-week, Open-label, Randomized, Multi-center, Parallel-group Study to Evaluate the Efficacy and Safety of Early Combination of Vildagliptin and Metformin in Patients With Type 2 Diabetes Mellitus Who Are Inadequately Controlled With Prior Metformin Monotherapy in Comparison to up Titrating Metformin Dose.
Brief Title: Galvus on Met Phase 4 Study : Study to Evaluate the Efficacy and Safety of Early Combination of Vildagliptin and Metformin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AKR03T
Record Dates: First submitted 2009-09-09; First posted 2009-09-11 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Galvus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; BID protein, human; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Galvus group (Experimental): the combination of metformin plus Vildagliptin:
  * vildagliptin 50 mg bid plus metformin 1500mg
  * Additional SU therapy(After 12th week only under the following conditions): If A1c is ≥ 7.0% or investigator determines that the patient have metabolic problems at 12th week of therapy, investigator can prescribe additional sulfonylurea(glimepiride) to the current therapy.
  Interventions: Drug: vildagliptin 50 mg bid plus metformin 1500mg (Galvus+Diabex)
- Diabex group (Active Comparator): metformin alone arm:
  * metformin 1500mg plus metformin 500mg or 1000mg
  * Additional SU therapy(After 12th week only under the following conditions): If A1c is ≥ 7.0% or investigator determines that the patient have metabolic problems at 12th week of therapy, investigator can prescribe additional sulfonylurea(glimepiride) to the current therapy
  Interventions: Drug: metformin 1500mg plus metformin 500mg or 1000mg (Diabex)

INTERVENTIONS:
Drug: vildagliptin 50 mg bid plus metformin 1500mg (Galvus+Diabex) — vildagliptin 50 mg bid plus metformin 1500mg
  Arms: Galvus group
Drug: metformin 1500mg plus metformin 500mg or 1000mg (Diabex) — metformin 1500mg plus metformin 500mg or 1000mg
  Arms: Diabex group

SUMMARY:
The study design of this trial is open-label, randomized, multi-center, parallel-group study.

DETAILED DESCRIPTION:
* The progressive nature of T2DM will require the use of combination therapy in many patients over time to achieve and maintain glycemic control. Early combination, compared with maximal dose of monotherapy, could be more effective in lowering glycemia with better tolerability.
* Vildagliptin is a new oral antidiabetic drug acting as a potent and selective inhibitor of dipeptidyl peptidase-4(DPP-4), the enzyme responsible for the rapid degradation of circulating glucagon-like peptide-1. Vildagliptin improves islet function by a mechanism of increasing plasma levels of the active forms of the incretin hormones, GLP-1 and GIP.
* Metformin improves hyperglycemia primarily through its suppression of hepatic gluconeogenesis as well as enhancement of peripheral glucose update. Metformin is the most commonly prescribed first-line antidiabetic drug worldwide, but due to the progressive worsening of blood glucose control during the natural history of type 2 diabetes, combination therapy usually becomes necessary.
* Thus their combination therapy with complimentary action mechanism could be as effective as up titration of monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus who were inadequately controlled (baseline A1c of 7.0~11.0%)on metformin monotherapy (1500mg metformin)for ≥ 2 months before baseline visit
* Age of 18-80 years
* Body Mass Index of 18-40 kg/m2

Exclusion Criteria:

* Type 1 of diabetes
* Myocardial Infarction, Unstable Angina, or Coronary Artery Bypass Graft within the previous 6 months
* Congestive Heart Failure (III or NYHA class IV)
* Liver disease such as cirrhosis or Chronic Active Hepatitis
* History of Lacticacidemia
* Use of any Oral Anti-diabetic Drug other than Metformin within the 2 months
* Use of insulin before screening visit
* ALT or AST >3 times the upper limit of Normal range
* Creatinine >1.5 mg/dl
* Other situation (pregnant or lactating females, history of drug or alcohol abuse, night-shift workers, clinically significant laboratory abnormality on screening or any medical condition that would affect the completion or outcome of the study)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c at 24 weeks | 32weeks

SECONDARY OUTCOMES:
Hemoglobin A1c at 12 weeks | 32weeks
Fasting plasma glucose(Self Monitored Blood Glucose) at 24 week | 32weeks
2hours post-prandial plasma glucose(Self Monitored Blood Glucose) at 24 week | 32weeks
Fasting Lipid profiles at 24 week | 32weeks
Body weight at 24 week | 32weeks
Hypoglycemic events, Gastro-Intestinal events, other adverse events at each visit | 32weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sei Hyun Baik, professor, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Handok Pharmaceuticals, Seoul, Seoul, South Korea